CLINICAL TRIAL: NCT00717119
Title: Evaluation of the Effect of the Association of Proton Pump Inhibitor (PPIs) With Non-Steriodal Anti-Inflamatories (NSAIDs) in Work Leave Time.
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Ibermutuamur M.A.T.E.P.S (Unknown)
Responsible Party: Mónica Tafalla/MD, PhD, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-GES-DUM-2008/3
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2008-09-15 (Estimated); Status verified 2008-07

CONDITIONS: Sprain of Ankle
Keywords: GI; NSAID; Complications; Treated; Patients
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with sprain of ankle treated with NSAID

SUMMARY:
Retrospective cohort study to evaluate the effect of the association of PPIs with NSAIDs in work leave time.

ELIGIBILITY:
Inclusion Criteria:

* Work leave due to a sprain of ankle

Exclusion Criteria:

* (none)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data base of patients with work leave due to a sprain of ankle
Sampling Method: Non-Probability Sample
Enrollment: 6356 (Actual)
Dates: Start 2008-04; Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Total work leave time | Jan 2007 to Dec 2007

SECONDARY OUTCOMES:
GI complications | Jan 2007 to Dec 2007
Direct medical costs | Jan 2007 to Dec 2007

CONTACTS AND LOCATIONS:
Overall Officials: Javier N Rivero, MSc, Study Director — Epidemiology Unit. AstraZeneca
Locations (1):
- Research Site, Madrid, Spain